CLINICAL TRIAL: NCT04271540
Title: Effects of Tildrakizumab on Coronary Microvascular Function in Moderate-Severe Psoriasis
Brief Title: MIcrovascular dysfuNction In Moderate-severe Psoriasis
Acronym: MINIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marcelo F. Di Carli, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Marcelo F. Di Carli, MD, FACC, Chief, Nuclear Medicine, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000200
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis; Cardiovascular Disease
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases | interventions — tildrakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Subjects treated with Tildrakizumab (Experimental): Informed consent will be obtained from study participants willing to participate in MiNIMA. Study participants will then undergo the baseline rest/stress cardiac PET scan. The final PET scan will occur at 6 months after the intervention.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — Tildrakizumab, a p19 inhibitor which blocks IL-23 and Th17 mediated inflammation, will be given for 6 months. As below, a baseline cardiac PET scan will be performed prior to initiation and after 6 months of treatment.
  Radiation: A cardiac PET scan will be performed at baseline and at 6 months
  Other Names: Ilumya

SUMMARY:
Psoriasis, a common chronic inflammatory skin disease affecting approximately 2% of the population, is associated with increased cardiovascular (CV) risk. Despite the implication of inflammation in this excess risk, it remains unclear whether reducing inflammation reduces the risk of cardiac events. This study proposes to test whether Tildrakizumab, an FDA approved therapy for psoriasis that blocks IL-23 and the Th17 pathway of inflammation, improves coronary vascular function and coronary flow reserve, as measured by noninvasive imaging with cardiac positron emission tomography. In so doing, improvement in coronary vasoreactivity, endothelial function, and tissue perfusion may have beneficial effects on myocardial mechanics, left ventricular deformation and function and, ultimately, symptoms and prognosis.

This research may offer novel insights into the contributors of CV risk in psoriasis and provide data to support the development of strategies to prevent cardiovascular events in psoriatic disease.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the impact of Tildrakizumab therapy on coronary vasoreactivity and myocardial mechanics, as indicators of subclinical cardiovascular disease in patients with psoriatic disease and intermediate-high CV risk. Impaired coronary flow reserve (CFR) is a measure of coronary vasoreactivity and a manifestation of myocardial ischemia which may precede clinical CV events (and visible changes in plaque morphology) in high-risk patients with psoriatic disease. From previous studies, it is known that traditional risk factors underestimate cardiovascular risk in psoriatic disease. Tildrakizumab, a p19 inhibitor which blocks IL-23 and Th17 mediated inflammation, is an FDA approved therapy for moderate-severe psoriasis and has been shown to reduce inflammation. Furthermore, IL-17 is associated with endothelial dysfunction and atherosclerosis. The central hypothesis is that reducing systemic inflammation using tildrakizumab will quantitatively improve myocardial blood flow and CFR as measured by PET over 6 months; and this improvement in coronary vasoreactivity, endothelial function, and tissue perfusion may have beneficial effects on myocardial mechanics, left ventricular function and, ultimately, symptoms and prognosis.

This is a single-arm open-label mechanistic clinical study in adult subjects with moderate-severe psoriasis and increased cardiovascular risk. We plan to enroll approximately 35 patients to receive Tildrakizumab over 6 months. The study will consist of 4-5 visits including a virtual or in person screening visit, a baseline visit in which baseline imaging tests will be conducted and study drug will be dispensed, two in person visits for which study drug will be given and monitoring of AE events and compliance, and a final visit in visit in which imaging tests will be repeated

ELIGIBILITY:
In order for an individual to participate, they must meet all of the inclusion and exclusion criteria as outlined below.

Inclusion Criteria include the following:

1. Moderate-to-severe psoriasis
2. Ages 18-90
3. Body surface area (BSA) involvement ≥ 3% OR 5-point Physician Global Assessment (PGA) Score ≥ 3 OR Psoriasis Area and Severity Index (PASI) score ≥ 12
4. Patients who have failed biologic therapy, topical steroids, phototherapy, or other systemic therapies will be required to have a wash-out period, which will be calculated accordingly to the specific drug (Appendix 1)
5. Evidence of at least one cardiovascular risk factor which includes hsCRP ≥ 2 mg/L, DM, obesity (BMI>25), hyperlipidemia, hypertension, family history of early coronary artery disease, or evidence of metabolic syndrome

   ---Metabolic syndrome defined as at least three of the following: glucose>100mg/dl or taking hypoglycemic agent, HDL<40mg/dl (men) or 50 mg/dl (women), triglycerides ≥150mg/dl, waist circumference >40 in mean or >35 in women, or blood pressure ≥130/85 or taking anti-hypertensive.
6. If the patient is on a statin therapy, they must be on a stable dose for at least 6 months prior to enrollment.

Exclusion Criteria include the following:

1. Documented history of other systemic inflammatory diseases, including SLE and RA, which in the opinion of the investigator would be inappropriate for enrollment.
2. Prior history of untreated chronic infection (tuberculosis), severe fungal infection, or known HIV positive, chronic hepatitis B or C infection), prior history of active solid malignancy, myeloproliferative or lymphoproliferative disease within 5 years, excluding treated non-melanoma skin cancer
3. Renal insufficiency (CrCl <40 ml/min)
4. NYHA class IV heart failure
5. Patients requiring chronic treatment with oral prednisone >10mg/day, methotrexate, or other immunosuppressive agents.
6. Pregnancy and Breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Di Carli, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects treated with Tildrakizumab
Started | 36
Completed | 30
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Screen Fail | 5

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Treated With Tildrakizumab
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Psoriasis Area and Severity Index (PASI) [Median (Inter-Quartile Range); unit: scores on a scale] — Psoriasis Area and Severity Index (PASI) is a measurement tool which assesses the severity of psoriasis. The range of absolute PASI scores is 0 to 72, with higher scores indicating a greater severity of psoriasis. A score of 0 indicates no psoriasis; a score of 0 to 5 indicates mild psoriasis; a score of 6 to 10 suggests moderate psoriasis; and a score of 11 or above suggests severe psoriasis.
  scores on a scale | 10.9 [6.7 to 15.6]
Physician's Global Assessment of Psoriasis (PGAP) [Median (Inter-Quartile Range); unit: scores on a scale] — Physician's Global Assessment of Psoriasis (PGAP) estimates a patient's overall severity of psoriasis at a given point in time. Psoriatic lesions are graded for induration, erythema, and scaling based on scales of 0 to 4 that are then averaged over all lesions. A score of 0 means no psoriasis, while a score of 4 indicates severe psoriasis.
  scores on a scale | 3.0 [2 to 3]
Number of Participants with Psoriatic Arthritis [Count of Participants; unit: Participants] | 10
Number of Participants with Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] — Participants with established CAD at baseline
  Participants | 5
Number of Participants with Hypertension [Count of Participants; unit: Participants] — Participants with established hypertension at baseline
  Participants | 17
Number of Participants with Diabetes mellitus [Count of Participants; unit: Participants] — Participants with established diabetes mellitus at baseline
  Participants | 5
Number of Participants with Obesity [Count of Participants; unit: Participants] — Participants with obesity at baseline, defined as BMI > 32
  Participants | 18
Number of Participants with Dyslipidemia [Count of Participants; unit: Participants] — Participants with dyslipidemia at baseline, as defined by screening lab or past medical history
  Participants | 24
Number of Participants with On Statin [Count of Participants; unit: Participants] — Participants on a statin at baseline
  Participants | 10
Atherosclerotic Coronary Artery Disease (ASCVD) Risk Score [Median (Inter-Quartile Range); unit: Percentage] — The 10 year Atherosclerotic Coronary Artery Disease (ASCVD) risk score was calculated using the ASCVD Risk Estimator by the American College of Cardiology. The risk score is a percentage, from 0-100%, estimating a patient's 10-year risk of having a heart attack or stroke. Risk scores of <10% are considered low, 10-<20% intermediate, and >=20% high.
  Percentage | 7 [4 to 23]
High-sensitivity Troponin T (Hs-TnT) [Median (Inter-Quartile Range); unit: mg/L] | 10 [6 to 24]
High-Sensitivity C-Reactive Protein (hs-CRP) [Median (Inter-Quartile Range); unit: mg/L] | 2.6 [0.3 to 60]
N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) [Median (Inter-Quartile Range); unit: pg/mL] | 57 [9 to 1425]
Lipid panel [Median (Inter-Quartile Range); unit: mg/dl] — Baseline standard lipid panel measurements
  mg/dl
    Total cholesterol | 191 [76 to 294]
    LDL | 103 [33 to 163]
    HDL | 50 [30 to 95]
    Triglycerides | 140 [45 to 339]
Coronary Flow Reserve (CFR) [Mean (Standard Deviation); unit: Ratio] — CFR is calculated as the ratio of peak hyperemic myocardial blood flow over that at rest
  Ratio | 2.63 (.72)
Myocardial Blood Flow (MBF) [Mean (Standard Deviation); unit: ml/min/g] — Quantified using myocardial perfusion Positron Emission Tomography (PET) imaging
  ml/min/g
    Global Rest MBF | 0.81 (.15)
    Global Stress MBF | 2.06 (.42)
CFR <2.5 [Count of Participants; unit: Participants] | 15
Heart rate (HR) [Mean (Standard Deviation); unit: bpm]
  Resting HR | 74 (31)
  Peak HR | 95.2 (27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Coronary Flow Reserve (CFR) After 6 Months of Therapy With Tildrakizumab
Description: Change (from baseline) in global CFR, as measured by PET imaging at 24 weeks after initiation of Tildrakizumab therapy.
  Coronary flow reserve (CFR), the ratio of peak vasodilator stress to rest myocardial blood flow (MBF), represents the maximal ability to augment coronary flow and myocardial perfusion. Absolute MBF was computed from the rest and stress myocardial perfusion PET images using commercially available software (Corridor4DM; Ann Arbor, Michigan) and a two-compartment tracer kinetic model. Impaired MBFR is defined as a ratio of <2.0, which is associated with increased cardiovascular risk.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: CFR Ratio
Arm/Group | Subjects treated with Tildrakizumab
Number analyzed (Participants) | 30
CFR Ratio | -0.03 (0.83)

2. Secondary Outcome: Correlation Between Change in Global CFR and Psoriasis Skin Severity
Description: Correlation between the change (from baseline) in global CFR and psoriasis skin severity scores (Body surface area [BSA], Physician's Global Assessment [PGA], Psoriasis Area and Severity Index [PASI]) at 24 weeks after initiation of Tildrakizumab
Time Frame: 24 weeks
Measure: Number; unit: Spearman's rank correlation coefficient
Arm/Group | Subjects treated with Tildrakizumab
Number analyzed (Participants) | 31
Spearman's rank correlation coefficient | 0.18
Statistical Analysis 1: Comparison: Subjects treated with Tildrakizumab; Test type: Superiority; p = 0.35, Spearman's Rank Correlation

3. Secondary Outcome: Change in Peak-stress Global Myocardial Blood Flow
Description: Change (from baseline) in peak-stress global myocardial blood flow (in mL/min/g) at 24 weeks after initiation of Tildrakizumab
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ml/min/g
Arm/Group | Subjects treated with Tildrakizumab
Number analyzed (Participants) | 30
ml/min/g | 0.07 (0.41)

4. Secondary Outcome: Change in Peak-stress Global Coronary Vascular Resistance
Description: Change (from baseline) in peak-stress global coronary vascular resistance (in mm Hg/mL/min/g) at 24 weeks after initiation of Tildrakizumab
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mm Hg/mL/min/g
Arm/Group | Subjects treated with Tildrakizumab
Number analyzed (Participants) | 30
mm Hg/mL/min/g | -1.1 (13.15)

ADVERSE EVENTS:
Time Frame: from enrollment until one week after completion of the trial, an average of 27 weeks
Arm/Group | Subjects treated with Tildrakizumab
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 3/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects treated with Tildrakizumab (N=31)
COVID infection (Infections and infestations) | 3

LIMITATIONS AND CAVEATS:
This study is a pilot, mechanistic study, and should be viewed in light of this. Larger studies are warranted with longer follow-up to address whether myocardial blood flow improves over a longer duration. Conversely, whether myocardial blood flow worsens in the absence of IL-23 blockade could only be examined in a patient population of moderate-severity who are not treated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04271540/Prot_SAP_000.pdf